CLINICAL TRIAL: NCT02579668
Title: Language Therapy in British Sign Language - a Pilot Study to Explore the Use of Therapeutic Strategies and Resources by Deaf Adults With Young People Who Have Language Difficulties in BSL.
Brief Title: Language Therapy in British Sign Language
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 13/0476
Record Dates: First submitted 2015-09-07; First posted 2015-10-19 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2015-10

CONDITIONS: Language Difficulties in British Sign Language
MeSH Terms: interventions — Language Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Language therapy in BSL (Experimental): Working with Deaf practitioners to provide language activities in British Sign Language aimed at developing children's language skills.
  Interventions: Other: Language Therapy

INTERVENTIONS:
Other: Language Therapy

SUMMARY:
In the United Kingdom, the language of the Deaf community is British Sign Language (BSL). A small proportion of Deaf young people who use BSL as their first or dominant language have specific language difficulties and would benefit from language therapy provided in sign language by adults who are fluent in BSL and may be Deaf. Some Deaf adults are currently employed in education and health services to support children's BSL development. However there is little training or information available to these adults about language assessment, diagnosis of language difficulties or intervention strategies.

Recent studies have highlighted language difficulties and therapy in sign as an issues and begun to explore Deaf adults understanding of language difficulties and disorder. This project aims to extend knowledge in this area by supporting Deaf practitioners to understand and develop language therapy skills and co-develop language therapy intervention resources. The study will pilot training for practitioners and language therapy interventions for young people.

DETAILED DESCRIPTION:
The study will be in three phases. The design has been discussed at regular Language Working Group Meetings with Deaf practitioner colleagues who may want to volunteer to be involved in the project.

In Phase 1, information will be sought from Deaf practitioners in focus groups and from questionnaires about the strategies and resources they currently employ when working with Deaf young people with language difficulties. This information will be compared to evidence based models of therapy for spoken English to see whether similar themes emerge. The findings will also be used to identify themes for other strategies and resources Deaf practitioners use which are not present in spoken English language therapy. The data gathered will be included in planning the next phase of the project. Scenarios and questions similar to those planned for the focus group and questionnaire have been trialed at Service training days and feedback has been gathered from staff involved.

Phase 2 will involve working with Deaf practitioners to develop and define strategies and resources for language therapy in BSL. These will be with a small group of three or four Deaf practitioners. Dynamic assessment and mediated learning principles will be used to identify key skills and resources for Deaf practitioners in providing language therapy.

This process, including pre and post involvement questionnaires, will use video observation and reflective practise tools. Analysis of a language therapy intervention session by a Deaf practitioner will provide a snapshot or 'assessment' of their initial skills and knowledge. Then, over a period of six sessions, videos of the Deaf practitioner working with a young person on language activities will be jointly analysed and reflected upon to identify strategies and resources that are or would be useful in this working context. This joint analysis between the researcher, a qualified Speech and Language Therapist, and the Deaf practitioner will provided teaching, learning and reflection opportunities. Finally the video analysis by the Deaf practitioner, without reflection with the researcher, will be repeated to give a second 'assessment' of the Deaf practitioner's skills and knowledge. The Deaf practitioner will be asked to give feedback on this process, identifying helpful strategies discussed, issues with the process and information they feel would be useful to other Deaf practitioners completing similar work with young people. Deaf practitioners will work with deaf young people who are currently on their clinical caseload and have previously been identified as having language difficulties. These young people and their families will be informed about the project and, if they consent to participate, will participate in the six sessions led by the Deaf practitioner.

The information gained from this process will identify useful strategies and resources. Validation will be sought by comparing evidence based language therapy strategies and resources from spoken English with those identified by Deaf practitioners in Phase 1 and those found to be useful by Deaf practitioners in Phase 2. These will be used to develop a training package containing strategies, resources and guiding principles for Deaf practitioners using BSL for language therapy delivery.

In phase 3, single case studies will be undertaken. These will include training other Deaf practitioners to use strategies and resources with Deaf young people. Qualitative information from Deaf practitioners and young people, as well as quantitative information from pre and post intervention language assessments and sample video clips, will be analysed to ascertain whether the training in strategies and resources enables Deaf practitioners to use identified intervention strategies and develop the language skills of Deaf young people. The qualitative data will be gathered through the use of reflective logs and questionnaires. The quantitative data will be gathered through the use of structured language assessment activities. Young people and their parents will also provide qualitative information about the process through questionnaires or interviews, depending on their communication mode (English, another spoken language or BSL) and their preference.

ELIGIBILITY:
Inclusion Criteria:

* National Deaf Child and AdolescentDeaf practitioners will be eligible to participate and only volunteers will be included that have manager's approval, are working with a young person who meets the inclusion criteria;
* Aged 8-15yrs
* Capacity to consent to participation in activities
* Language difficulties in BSL identified in their care plan
* Consent from carers/parents

Exclusion Criteria:

* Young people with a diagnosis of Autism Spectrum Disorder, severe mental illness of risk factors that would make intervention unsafe.

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Qualitative questionnaire measure of Deaf participants views. | Up to ten months
  Deaf practitioners will provide their views on how training and supervision for intervention activities has impacted on their skills and understanding.